CLINICAL TRIAL: NCT05342025
Title: Investigation Of The Effects Of Proprioceptive Neuromuscular Facilitation Techniques For Upper Extremity And Trunk, Combined With Respiration, On Respiratory Capacity And Swallowing In Individuals With Multiple Sclerosis
Brief Title: Proprioceptive Neuromuscular Facilitation in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Assoc.Prof. Dr., Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-KAEK-57-21-02
Record Dates: First submitted 2022-04-14; First posted 2022-04-22 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Multiple Sclerosis
Keywords: respiratory function; swallowing; proprioceptive neuromuscular facilitation
MeSH Terms: conditions — Multiple Sclerosis; Respiratory Aspiration | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessor will be blind to the randomization and the investigator will be blind to the results of the assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF group (Experimental): PNF will be applied to the trunk and upper extremities combined with breathing, 3 times a week, 1 hour a day for 6 weeks. The physiotherapist will apply pressure and stretches to the chest wall and diaphragm for 20 seconds by giving verbal commands to the patient for the inspiration/expiratory phases. The physiotherapist will apply patterns over the 2nd and 3rd ribs in a bilateral anterior manner including intercostal stretches.
  Interventions: Other: PNF
- Control Group (Active Comparator): Individuals in this group will be taught breathing exercises (diaphragmatic breathing, thoracic expansion, pursed-lip breathing, and respiratory control) after the assessments, and they will be informed about performing breathing exercises for 15 minutes a day, every day of the week. Patients will be asked to keep a "treatment diary" to control regular breathing exercises. Individuals will be re-evaluated after 2 months.
  Interventions: Other: Breathing exercises

INTERVENTIONS:
Other: PNF — PNF will be applied to the trunk and upper extremities combined with breathing, 3 times a week, 1 hour a day for 6 weeks. Breathing PNF patterns, pressure, and stretches will be applied inward and upwards into the rib cage so that they do not cause pain. Diaphragmatic stimulation will be performed on both sides with repeated contractions, hand contacts, and stabilization techniques. Facilitation techniques will be used to stimulate the intrinsic respiratory muscles. Again, with respect to inspiration, the patterns will be studied in neck extension, upper and lower trunk extension, and upper extremities flexion patterns. Neck flexion, upper and lower trunk flexion, and extension patterns of the upper extremities will be applied in relation to expiration. The physiotherapist will apply pressure and stretches to the chest wall and diaphragm for 20 seconds by giving verbal commands to the patient for the inspiration/expiratory phases.
  Arms: PNF group
Other: Breathing exercises — Breathing exercises: diaphragmatic breathing, thoracic expansion, pursed-lip breathing and respiratory control for 15 minutes a day, every day of the week.
  Arms: Control Group

SUMMARY:
Multiple Sclerosis (MS) is an autoimmune central nervous system disease characterized by inflammation, demyelination, and axonal degeneration. Clinical symptoms of the disease include fatigue, speech, breathing, and swallowing problems. Although respiratory issues are less common in patients with MS, pulmonary complications are among the most common causes of mortality and morbidity in the terminal period. Although it is known that expiratory and inspiratory respiratory muscle training is beneficial in MS disease, the protocols used are variable and there is no standard exercise protocol. Respiratory muscle training is one of the instrument-oriented techniques, and the issue of delivering these devices to each patient creates a cost disadvantage. It is foreseen that the preference for the PNF technique to be applied in combination with respiration in the project will enable the development of alternative treatment approaches in order to solve the researched problems in MS disease, which is a critical health problem. Proprioceptive Neuromuscular Facilitation (PNF) is defined as facilitating the responses of the neuromuscular mechanism by stimulating the proprioceptors. In the literature, there is no study examining the effectiveness of PNF on respiratory and swallowing functions in individuals with MS. The aim of the study is to investigate the effects of PNF application in combination with upper extremity and trunk patterns on respiratory and swallowing functions in patients with MS.

DETAILED DESCRIPTION:
Among the physiotherapy and rehabilitation approaches applied for the problems affecting the quality of life in Multiple Sclerosis; Exercises for muscle strength loss, balance coordination exercises, electrical stimulation, orthotic approaches, breathing and swallowing exercises, and Proprioceptive Neuromuscular Facilitation (PNF) techniques are included. Among the respiratory dysfunctions are seen in MS patients: abnormal respiratory control, respiratory muscle weakness, bulbar dysfunction/respiratory failure, and sleep breathing disorders can be cited as examples. Significant expiratory weakness develops in MS patients with the progression of the disease, and the accompanying upper extremity involvement exacerbates this problem. It should not be ignored that swallowing-respiratory coordination and ultimately swallowing can be affected by the deterioration of respiration in MS patients. Among the neurophysiological approaches, the PNF technique; is known to have positive effects on tidal volume, respiratory rate, and minute ventilation parameters in neurological patients. Respiratory patterns of PNF can be applied alone or in combination with other extremity patterns. This study aims to examine the effect of using PNF breathing techniques in combination with upper extremity and trunk on MS patients on respiratory and swallowing functions.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 25-55,
* MS was diagnosed by a neurologist,
* Expanded Disability Status Scale (EDSS) - Expanded Disability Status Scale (EDSS) score between 1-5,
* Have not had an attack in the last 3 months,
* Have not participated in any respiratory-based physiotherapy and rehabilitation program in the last 6 months,
* Not having orthopedic problems, persistent neck pain and/or radiculopathy that would prevent them from participating in the study,
* Individuals willing to participate in the study will be included.

Exclusion Criteria:

* Having chest wall deformity,
* Having chronic cardiac or pulmonary disease such as COPD, asthma, interstitial lung disease and heart failure that may affect respiratory muscle strength and respiratory functions,
* Having pneumonia due to viral or bacterial infection in the last 6 months,
* Having COVID-19,
* Having a diagnosed psychiatric disorder,
* Using tobacco and tobacco products,
* Individuals with cooperation problems that may hinder assessments and treatment will not be included.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume 1st second | 8 weeks
  Spirometric assessment will be performed to determine participants' forced expiratory volume in one second (FEV1).
Peak cough flow | 8 weeks
  Peak cough flow (PEF) will be measured in triplicate during the "maximal coughing manoeuvre" with a digital PEFmeter.
Respiratory muscle strength | 8 weeks
  The respiratory muscle strength measurement of the participants will be made with an intraoral pressure measuring device, an intraoral pressure gauge. Maximal inspiratory and expiratory pressures will be measured.
Forced vital capacity | 8 weeks
  Spirometric assessment will be performed to determine participants' forced vital capacity (FVC).

SECONDARY OUTCOMES:
2 Minutes Walking Test | 8 weeks
  The 2 Minute Walk Test (2MWT) is a measure of self-paced walking ability and functional capacity[1], particularly for those who cannot manage the longer Six Minute Walk Test (6MWT) or 12 Minute Walk Test.
Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL) | 8 weeks
  It is a disease-specific quality of life scale and consists of a total of 31 questions, including 3 subheadings: psychological, physical and psychosocial.
Eating Assessment Tool (EAT-10) | 8 weeks
  It is used to evaluate dysphagia symptom severity and response to treatment. The single-factor scale consists of 10 items scored between 0-4.
Fatigue Severity Scale (Fatigue Severity Scale) | 8 weeks
  The scale consists of 9 questions that evaluate fatigue and are scored between 1-7. High scores indicate increased fatigue.
Dysphagia Rating Scale in Multiple Sclerosis (DYMUS) | 8 weeks
  The scale is used in the evaluation of oropharyngeal dysphagia in patients with MS.DYMUS is a 10-item questionnaire; all the answers are dichotomous, coded as 1 or 0, depending on the presence or the absence of the event

CONTACTS AND LOCATIONS:
Overall Officials: Buket AKINCI, Assoc.Prof., Study Chair — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No